CLINICAL TRIAL: NCT01553903
Title: Feasibility Study for the Determination of Oxysterols in Patients With Breast Cancer Receiving Hormonal Therapy With Tamoxifen or Not
Acronym: OXYTAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11 SEIN 09
Record Dates: First submitted 2011-12-20; First posted 2012-03-14 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
Keywords: Hormonal therapy; Breast Cancer; AEBS; Oxysterols
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; exemestane; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tamoxifen, (Experimental): Current hormonotherapy treatment in hormone dependent breast cancer
  Interventions: Drug: Tamoxifen,
- Exemestane (Experimental): Current hormonotherapy treatment in hormone dependent breast cancer
  Interventions: Drug: Exemestane
- Anastrozole (Experimental): Current hormonotherapy treatment in hormone dependent breast cancer
  Interventions: Drug: Anastrozole
- Letrozole (Experimental): Current hormonotherapy treatment in hormone dependent breast cancer
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Tamoxifen, — Tamoxifen 20 mg/day during 5 years,
  Arms: Tamoxifen,
Drug: Exemestane — Exemestane 25mg/day during 5 years
  Arms: Exemestane
Drug: Anastrozole — Anastrozole 1 mg/day during 5 years,
  Arms: Anastrozole
Drug: Letrozole — Letrozole 2.5 mg/day during 5 years,
  Arms: Letrozole

SUMMARY:
This is a biomedical study of interventional type which includes 29 patients on 9 months: 8 months recruiting and 1 month follow up.

Patients with hormone dependent breast cancer metastatic or non-metastatic, for which an indication of hormonal therapy treatment (with tamoxifen or anti-aromatase) is retained, will be enrolled in this study.

The main objective of this study is to evaluate the feasibility for the determination of Oxysterols (CT, CE, OCDO) in this patient population, before and after the initiation of treatment (ie, at D0 before and D28 after beginning of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Women of more than 18 years old (menopause or not).
2. Women with invasive breast cancer metastatic or non-metastatic, for which treatment with tamoxifen or anti-aromatase is retained.
3. Cancer hormone-expressing estrogen receptor (ER) and / or progesterone receptor (PR) (≥ 10% of tumor cells in Technical HIC).
4. Any previous hormonal therapy, stopped for progression, should be discontinued for at least 21 days prior to study entry.
5. WHO ≤ 2.
6. Women of childbearing age must use effective contraception for the duration of the study.
7. Informed consent obtained and signed before any specific procedure in the study.
8. Patient member in a national insurance scheme.

Exclusion Criteria:

1. Patient with breast cancer HER2 positive (IHC and / or FISH-CISH)
2. Patient already receiving hormonal therapy or patient who has not stopped hormonal therapy for at least 21 days.
3. Patient that should receive a chemotherapy and / or another targeted therapy (other than hormonal therapy) for the treatment of the breast cancer.
4. Any other medical or psychiatric condition or laboratory abnormality severe, acute or chronic making the inclusion of the patient in the study inappropriate in the opinion of the investigator.
5. Patient unable to follow procedures, visits, examinations described in the study.
6. Pregnant women or nursing mothers can not participate in the study.
7. Patients under legal guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Determination of Oxysterols (OCDO, CT and CE)plasma concentrations by Gaz Chromatography coupled to mass spectrometry (GC/MS)in human. | 2 time points (D0 and D28) over a period of 2 years
  Oxysterols measured are the following : OCDO (6-oxo-cholestan-3 beta, 5 alpha-diol), CE (cholesterol-5,6-eposides) and CT (cholestane-3 beta, 5 alpha, 6 beta-triol).
  Calibration curve will be established for each Oxysterol by GC/MS using deuterated analogues of each oxysterols for the quantification.

SECONDARY OUTCOMES:
Measure of Oxysterols (OCDO, CT and CE) plasma concentrations in patient treated with Tamoxifen | 2 time points (D0 and D28) over a period of 2 years
  Plasma concentrations of Oxysterols evaluated by Gaz chromatography coupled to mass spectrometry (GC/MS)in patients after 28 days of hormonal therapy with Tamoxifen in order to determine the impact of the treatment on these plasmatic concentrations(D28 oxysterols plasma concentrations will be compared to D0 oxysterols plasma concentrations)
Measure of Oxysterols (OCDO, CT and CE) plasma concentrations in patient treated with anti-aromatase. | 2 time points (D0 and D28) over a period of 2 years
  Plasma concentrations of Oxysterols evaluated by Gaz chromatography coupled to mass spectrometry (GC/MS)in patients after 28 days of hormonal therapy with anti-aromatase (Anastrozole, Letrozole or Exemestane) in order to determine the absence of impact of the treatment on these plasmatic concentrations (D28 oxysterols plasma concentrations will be compared to D0 oxysterols plasma concentrations).

CONTACTS AND LOCATIONS:
Overall Officials: Florence DALENC, MD, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius REGAUD, Toulouse, France